CLINICAL TRIAL: NCT02410772
Title: Rifapentine-containing Treatment Shortening Regimens for Pulmonary Tuberculosis: A Randomized, Open-label, Controlled Phase 3 Clinical Trial. TBTC Study 31, ACTG Study A5349
Brief Title: TBTC Study 31: Rifapentine-containing Tuberculosis Treatment Shortening Regimens
Acronym: S31/A5349
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6655
Record Dates: First submitted 2015-02-08; First posted 2015-04-08 (Estimated); Results first posted 2021-09-28 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — rifapentine; Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Regimen 1 (Active Comparator): Eight weeks of daily treatment with rifampin, isoniazid, pyrazinamide, and ethambutol, followed by Eighteen weeks of daily treatment with rifampin and isoniazid
  All drugs are administered orally, seven days/week, directly observed by a health care worker at least five of the seven days each week. Pyridoxine (vitamin B6), 25 or 50 mg, is administered with each study dose.
  study drug doses: rifampin, 600 mg; isoniazid, 300 mg; pyrazinamide, < 55kg 1000 mg, >= 55-75 kg 1500 mg, >75 kg 2000 mg; ethambutol, < 55kg 800 mg, >= 55-75 kg 1200 mg, >75 kg 1600 mg
  Interventions: Drug: control
- Regimen 2 (Experimental): Eight weeks of daily treatment with rifapentine, isoniazid, pyrazinamide, and ethambutol, followed by Nine weeks of daily treatment with rifapentine and isoniazid
  All drugs are administered orally, seven days/week, directly observed by a health care worker at least five of the seven days each week. Pyridoxine (vitamin B6), 25 or 50 mg, is administered with each study dose.
  study drug doses: rifapentine 1200 mg; isoniazid, 300 mg; pyrazinamide, < 55kg 1000 mg, >= 55-75 kg 1500 mg, >75 kg 2000 mg; ethambutol, < 55kg 800 mg, >= 55-75 kg 1200 mg, >75 kg 1600 mg
  Interventions: Drug: rifapentine
- Regimen 3 (Experimental): Eight weeks of daily treatment with rifapentine, isoniazid, pyrazinamide, and moxifloxacin, followed by Nine weeks of daily treatment with rifapentine, isoniazid, and moxifloxacin
  All drugs are administered orally, seven days/week, directly observed by a health care worker at least five of the seven days each week. Pyridoxine (vitamin B6), 25 or 50 mg, is administered with each study dose.
  study drug doses: rifapentine 1200 mg; isoniazid, 300 mg; pyrazinamide, < 55kg 1000 mg, >= 55-75 kg 1500 mg, >75 kg 2000 mg; moxifloxacin, 400 mg
  Interventions: Drug: rifapentine and moxifloxacin

INTERVENTIONS:
Drug: rifapentine — Regimen 2: Rifapentine is substituted for rifampin as the basis of 4-month treatment
  Other Names: Priftin
  Arms: Regimen 2
Drug: rifapentine and moxifloxacin — Regimen 3: In addition to the single substitution described for regimen 2, a second substitution is added, of moxifloxacin for ethambutol.
  Other Names: Priftin and Avelox
  Arms: Regimen 3
Drug: control — standard six-month treatment
  Arms: Regimen 1

SUMMARY:
The purpose of this study is to determine whether one or two four-month regimens of tuberculosis treatment are as effective as a standard six-month regimen for treatment of pulmonary tuberculosis (TB). All three regimens are administered daily, seven days each week, with direct observation of each dose by a health-care worker at least five of the seven days of each week.

The standard six-month regimen is two months of isoniazid, rifampin, ethambutol, and pyrazinamide followed by four months of isoniazid and rifampin.

The first short regimen is a single substitution of rifapentine for rifampin: two months of isoniazid, rifapentine, ethambutol, and pyrazinamide, followed by two months of isoniazid and rifapentine.

The second short regimen is a double substitution of rifapentine for rifampin and moxifloxacin for ethambutol: two months of isoniazid, rifapentine, moxifloxacin, and pyrazinamide, followed by two months of isoniazid, rifapentine, and moxifloxacin.

Target enrollment is 2500 participants. Each study participant will remain in the study for 18 months in order to include at least 12 months of evaluation of whether the participant's TB recurs.

DETAILED DESCRIPTION:
Title:

Rifapentine-containing treatment shortening regimens for pulmonary tuberculosis: a randomized, open-label, controlled, phase 3 clinical trial

Hypotheses:

A) Seventeen (17) week rifapentine-based regimen In previously untreated individuals with active drug-susceptible pulmonary tuberculosis treated with eight weeks of rifapentine (P), isoniazid (H), pyrazinamide (Z) and ethambutol (E) followed by nine weeks of rifapentine plus isoniazid, all given daily throughout, the proportion of participants who experience absence of cure (unfavorable outcome) will not be inferior to that observed in participants who are treated with a standard regimen (eight weeks of rifampin (R), isoniazid, pyrazinamide and ethambutol followed by eighteen weeks of rifampin plus isoniazid), all given daily throughout.

B) Seventeen (17) week rifapentine- plus moxifloxacin-containing regimen In previously untreated individuals with active drug-susceptible pulmonary tuberculosis treated with eight weeks of rifapentine, isoniazid, pyrazinamide and moxifloxacin (M), followed by nine weeks of rifapentine, isoniazid, and moxifloxacin, all given daily throughout, the proportion of participants who experience absence of cure (unfavorable outcome) will not be inferior to that observed in participants who are treated with a standard regimen (eight weeks of rifampin, isoniazid, pyrazinamide and ethambutol followed by eighteen weeks of rifampin plus isoniazid), all given daily throughout.

Phase: 3

Design: This will be an international, multicenter, randomized, controlled, open-label, 3-arm, phase 3 non-inferiority trial.

Population: Patients with newly diagnosed, previously untreated pulmonary tuberculosis.

Number of Sites: Multiple international sites, primarily sites of the Tuberculosis Trials Consortium and the AIDS Clinical Trials Group.

Study Duration: Duration per participant is approximately 18 months.

Description of Agent or Intervention: After written informed consent, participants will be randomly assigned to receive one of the following oral regimens:

Regimen 1 (control regimen): 2RHZE/4RH

* Eight weeks of daily treatment with rifampin, isoniazid, pyrazinamide, and ethambutol, followed by
* Eighteen weeks of daily treatment with rifampin and isoniazid

Regimen 2 (investigational regimen): 2PHZE/2PH

* Eight weeks of daily treatment with rifapentine, isoniazid, pyrazinamide, and ethambutol, followed by
* Nine weeks of daily treatment with rifapentine and isoniazid

Regimen 3 (investigational regimen): 2PHZM/2PHM

* Eight weeks of daily treatment with rifapentine, isoniazid, pyrazinamide, and moxifloxacin, followed by
* Nine weeks of daily treatment with rifapentine, isoniazid, and moxifloxacin

Objectives:

Primary:

* To evaluate the efficacy of a rifapentine-containing regimen to determine whether the single substitution of rifapentine for rifampin makes it possible to reduce to seventeen weeks the duration of treatment for drug-susceptible pulmonary tuberculosis
* To evaluate the efficacy of a rifapentine-containing regimen that in addition substitutes moxifloxacin for ethambutol and continues moxifloxacin during the continuation phase to determine whether it is possible to reduce to seventeen weeks the duration of treatment for drug-susceptible pulmonary tuberculosis

Secondary:

* To evaluate the safety of the investigational regimens
* To evaluate the tolerability of the investigational regimens
* To collect and store biospecimens from consenting participants for the purpose of future research on discovery and validation of TB biomarkers
* To determine the correlation of mycobacterial and clinical markers with time to culture conversion, culture status at completion of eight weeks of treatment, treatment failure, and relapse.
* To conduct a pharmacokinetic/pharmacodynamic (PK/PD) study of the test drugs. The main objectives of the PK/PD study are to characterize study drug PK parameters and to determine relationships between treatment outcomes and PK parameters.
* To evaluate the pharmacokinetics of efavirenz-based antiretroviral treatment among patients with TB/HIV co-infection taking efavirenz-based combination antiretroviral therapy and TB treatment with rifapentine

Endpoints:

Primary Endpoints:

* Efficacy: TB disease-free survival at twelve months after study treatment assignment.
* Safety: Proportion of participants with grade 3 or higher adverse events during study drug treatment

Secondary Endpoints:

* TB disease-free survival at eighteen months after study treatment assignment
* Time to stable sputum culture conversion (solid and liquid media considered separately)
* Speed of decline of sputum viable bacilli by automated liquid MGIT culture days to detection
* Proportion of participants who are culture negative at completion of eight weeks of treatment (solid and liquid media considered separately)
* Sensitivity analyses assuming all participants classified as 'not assessable' have a favorable outcome
* Discontinuation of assigned treatment for a reason other than microbiological ineligibility
* Estimated steady state efavirenz PK parameters including mid-dosing interval concentration

ELIGIBILITY:
Inclusion Criteria:

* Suspected pulmonary tuberculosis plus one or both of the following: a) at least one sputum specimen positive for acid-fast bacilli on smear microscopy OR b) at least one sputum specimen positive for M. tuberculosis by Xpert MTB/RIF testing, with semiquantitative result of 'medium' or 'high' and rifamycin resistance not detected.
* Age twelve (12) years or older
* A verifiable address or residence location that is readily accessible for visiting, and willingness to inform the study team of any change of address during the treatment and follow-up period.
* Women of child-bearing potential who are not surgically sterilized must agree to practice a barrier method of contraception or abstain from heterosexual intercourse during study drug treatment.
* Documentation of HIV infection status.
* For HIV-positive individuals, CD4 T cell count greater than or equal to 100 cells/mm3 based on testing performed at or within 30 days prior to screening.
* Laboratory parameters done at or within 14 days prior to screening:

  * Serum or plasma alanine aminotransferase (ALT) less than or equal to 3 times the upper limit of normal
  * Serum or plasma total bilirubin less than or equal to 2.5 times the upper limit of normal
  * Serum or plasma creatinine level less than or equal to 2 times the upper limit of normal
  * Serum or plasma potassium level greater than or equal to 3.5 meq/L
  * Hemoglobin level of 7.0 g/dL or greater
  * Platelet count of 100,000/mm3 or greater
* For women of childbearing potential, a negative pregnancy test at or within seven (7) days prior to screening
* Karnofsky score greater than or equal to 60
* Written informed consent

Exclusion Criteria:

* Pregnant or breast-feeding.
* Unable to take oral medications.
* Previously enrolled in this study.
* Received any investigational drug in the past 3 months.
* More than five (5) days of treatment directed against active tuberculosis within 6 months preceding initiation of study drugs.
* More than five (5) days of systemic treatment with any one or more of the following drugs within 30 days preceding initiation of study drugs: isoniazid, rifampin, rifabutin, rifapentine, ethambutol, pyrazinamide, kanamycin, amikacin, streptomycin, capreomycin, moxifloxacin, levofloxacin, gatifloxacin, ofloxacin, ciprofloxacin, other fluoroquinolones, ethionamide, prothionamide, cycloserine, terizidone, para-aminosalicylic acid, linezolid, clofazimine, delamanid or bedaquiline.
* Known history of prolonged QT syndrome.
* Suspected or documented tuberculosis involving the central nervous system and/or bones and/or joints, and/or miliary tuberculosis and/or pericardial tuberculosis.
* Current or planned use within six months following enrollment of one or more of the following medications: HIV protease inhibitors, HIV integrase inhibitors, HIV entry and fusion inhibitors, HIV non-nucleoside reverse transcriptase inhibitors other than efavirenz, quinidine, procainamide, amiodarone, sotalol, disopyramide, ziprasidone, or terfenadine. Individuals who are currently taking efavirenz-based antiretroviral treatment or for whom initiation of efavirenz-based antiretroviral treatment is planned within 17 weeks following enrollment may participate.
* Weight less than 40.0 kg.
* Known allergy or intolerance to any of the study medications.
* Individuals will be excluded from enrollment if, at the time of enrollment, their M. tuberculosis isolate is already known to be resistant to any one or more of the following: rifampin, isoniazid, pyrazinamide, ethambutol, or fluoroquinolones.
* Other medical conditions, that, in the investigator's judgment, make study participation not in the individual's best interest.
* Current or planned incarceration or other involuntary detention.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2516 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2021-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Dorman, MD, Study Chair — Medical University of South Carolina; Payam Nahid, MD, MPH, Study Chair — University of California at San Francisco; Susan Swindells, MBBS, Study Chair — University of Nebraska; Richard Chaisson, MD, Study Chair — Johns Hopkins University; Ekaterina V Kurbatova, MD, PhD, MPH, Study Chair — Centers for Disease Control and Prevention
Locations (33):
- United States (5):
  - TBTC Site 82/ ACTG Site 801 USCF AIDS CRS, San Francisco, California
  - TBTC Site 24 Columbia Unversity, New York, New York
  - TBTC Site 20 UNTHSC (University of North Texas Health Science Center), Fort Worth, Texas
  - TBTC Site 62 Baylor College of Medicine & Affiliated Hospitals/VA, Houston, Texas
  - TBTC Site 63 San Antonio VA Medical Center (South Texas Group), San Antonio, Texas
- Brazil (2):
  - TBTC Site 94/ ACTG Site 12201 Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - TBTC Site 91/ ACTG Site 12101 Insituto Nacional de Pesquisa Clínica Evandro Chagas, Rio de Janeiro
- TBTC Site 36 TB and Chest Service of Hong Kong, China, Hong Kong, China
- Haiti (2):
  - TBTC Site 67/ ACTG Site 31730 GHESKIO centers IMIS, Port-au-Prince, Ouest
  - TBTC Site 45/ ACTG Site 30022: Les Centres Gheskio (INLR), Port-au-Prince, Ouest
- India (2):
  - TBTC Site 43/ ACTG Site 31441 BJ Medical College, Pune, Maharashtra
  - TBTC Site 44/ ACTG Site 11701 CART CRS, YRGCARE Medical Centre VHS, Chennai, Tamil Nadu
- Kenya (3):
  - TBTC Site 02/ ACTG 12501 Kenya Medical Research Institute/Walter Reed Project Clinical Research Center (KEMRI/WRP) CRS, Kericho, Kericho County
  - TBTC Site 39/ ACTG Site 31460 Kisumu CRS, Kisumu, Nyanza Province
  - TBTC Site 03/ ACTG Site 12601 Moi University Clinical Research Site, Eldoret
- Malawi (2):
  - TBTC Site 04/ ACTG Site 30301 Blantyre CRS (or College of Medicine - Johns Hopkins Research Project, COM-JHP), Blantyre
  - TBTC Site 05/ ACTG Site 12001 UNC Project Tidziwe Centre, Lilongwe
- Peru (2):
  - TBTC Site 90/ ACTG Site 11301 Asociacion Civil Impacta Salud y Educacion, Lima
  - TBTC Site 93/ ACTG Site 11302 CRS San Miguel, Lima
- South Africa (8):
  - TBTC Site 10/ ACTG Site 31718 TASK Applied Science, Bellville, Cape Town
  - TBTC Site 09/ ACTG Site 31792 University of Cape Town Lung Institute (Pty) Ltd, Mowbray, Cape Town
  - TBTC Site 34 Wits Health Consortium Perinatal HIV Research Unit (PHRU), Soweto, Gauteng
  - TBTC Site 49/ ACTG Site 12301 Soweto ACTG CRS, Soweto, Johannesburg
  - TBTC Site 06/ ACTG Site 11201 Durban International Clinical Research Site, Durban, KwaZulu-Natal
  - TBTC Site 01/ACTG Site 8950 FAM CRU, Parow Valley, Western Cape
  - TBTC Site 08/ ACTG Site 31793 South African Tuberculosis Vaccine Initiative (SATVI), Cape Town, Western Province
  - TBTC Site 07/ ACTG Site 11101 Wits Helen Joseph CRS, Johannesburg
- Thailand (2):
  - TBTC Site 42/ ACTG Site 31802 The Thai Red Cross AIDS Research Centre, Pathumwan, Bangkok
  - TBTC Site 69/ ACTG Site 31784 Thai-CTIU, CMU HIV Treatment CRS, Muang Chiang Mai, Chiang Mai
- Uganda (2):
  - TBTC Site 11/ ACTG Site 12401 Joint Clinical Research Centre, Kampala Clinical Research Site, Kampala
  - TBTC Site 30 Uganda-Case Western Reserve Research Collaboration, Kampala
- TBTC Site 37 Vietnam NTP/UCSF Research Collaboration, Hanoi, Vietnam
- TBTC Site 41/ ACTG Site 30313 Parirenyatwa Clinical Research Site, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
Data being collected in CDISC format.

REFERENCES:
- [Derived] Chang VK, Imperial MZ, Phillips PPJ, Velasquez GE, Nahid P, Vernon A, Kurbatova EV, Swindells S, Chaisson RE, Dorman SE, Johnson JL, Weiner M, Jindani A, Harrison T, Sizemore EE, Whitworth W, Carr W, Bryant KE, Burton D, Dooley KE, Engle M, Nsubuga P, Diacon AH, Nhung NV, Dawson R, Savic RM; AIDS Clinical Trial Group; Tuberculosis Trials Consortium. Risk-stratified treatment for drug-susceptible pulmonary tuberculosis. Nat Commun. 2024 Oct 30;15(1):9400. doi: 10.1038/s41467-024-53273-7. PMID 39477924
- [Derived] Xu AY, Velasquez GE, Zhang N, Chang VK, Phillips PPJ, Nahid P, Dorman SE, Kurbatova EV, Whitworth WC, Sizemore E, Bryant K, Carr W, Brown NE, Engle ML, Nhung NV, Nsubuga P, Diacon A, Dooley KE, Chaisson RE, Swindells S, Savic RM. Pyrazinamide Safety, Efficacy, and Dosing for Treating Drug-Susceptible Pulmonary Tuberculosis: A Phase 3, Randomized Controlled Clinical Trial. Am J Respir Crit Care Med. 2024 Dec 1;210(11):1358-1369. doi: 10.1164/rccm.202401-0165OC. PMID 39012226
- [Derived] Ngo HX, Xu AY, Velasquez GE, Zhang N, Chang VK, Kurbatova EV, Whitworth WC, Sizemore E, Bryant K, Carr W, Weiner M, Dooley KE, Engle M, Dorman SE, Nahid P, Swindells S, Chaisson RE, Nsubuga P, Lourens M, Dawson R, Savic RM. Pharmacokinetic-Pharmacodynamic Evidence From a Phase 3 Trial to Support Flat-Dosing of Rifampicin for Tuberculosis. Clin Infect Dis. 2024 Jun 14;78(6):1680-1689. doi: 10.1093/cid/ciae119. PMID 38462673
- [Derived] Kurbatova EV, Phillips PPJ, Dorman SE, Sizemore EE, Bryant KE, Purfield AE, Ricaldi J, Brown NE, Johnson JL, Wallis CL, Akol JP, Ocheretina O, Van Hung N, Mayanja-Kizza H, Lourens M, Dawson R, Nhung NV, Pierre S, Musodza Y, Shenje J, Badal-Faesen S, Vilbrun SC, Waja Z, Peddareddy L, Scott NA, Yuan Y, Goldberg SV, Swindells S, Chaisson RE, Nahid P. A Standardized Approach for Collection of Objective Data to Support Outcome Determination for Late-Phase Tuberculosis Clinical Trials. Am J Respir Crit Care Med. 2023 May 15;207(10):1376-1382. doi: 10.1164/rccm.202206-1118OC. PMID 36790881
- [Derived] Pettit AC, Phillips PPJ, Kurbatova E, Vernon A, Nahid P, Dawson R, Dooley KE, Sanne I, Waja Z, Mohapi L, Podany AT, Samaneka W, Savic RM, Johnson JL, Muzanyi G, Lalloo UG, Bryant K, Sizemore E, Scott N, Dorman SE, Chaisson RE, Swindells S; Tuberculosis Trials Consortium (TBTC) Study 31/AIDS Clinical Trials Group (ACTG) A5349 study team. Rifapentine With and Without Moxifloxacin for Pulmonary Tuberculosis in People With Human Immunodeficiency Virus (S31/A5349). Clin Infect Dis. 2023 Feb 8;76(3):e580-e589. doi: 10.1093/cid/ciac707. PMID 36041016
- [Derived] Podany AT, Pham M, Sizemore E, Martinson N, Samaneka W, Mohapi L, Badal-Faesen S, Dawson R, Johnson JL, Mayanja H, Lalloo U, Whitworth WC, Pettit A, Campbell K, Phillips PPJ, Bryant K, Scott N, Vernon A, Kurbatova EV, Chaisson RE, Dorman SE, Nahid P, Swindells S, Dooley KE, Fletcher CV. Efavirenz Pharmacokinetics and Human Immunodeficiency Virus Type 1 (HIV-1) Viral Suppression Among Patients Receiving Tuberculosis Treatment Containing Daily High-Dose Rifapentine. Clin Infect Dis. 2022 Sep 10;75(4):560-566. doi: 10.1093/cid/ciab1037. PMID 34918028
- [Derived] Dorman SE, Nahid P, Kurbatova EV, Phillips PPJ, Bryant K, Dooley KE, Engle M, Goldberg SV, Phan HTT, Hakim J, Johnson JL, Lourens M, Martinson NA, Muzanyi G, Narunsky K, Nerette S, Nguyen NV, Pham TH, Pierre S, Purfield AE, Samaneka W, Savic RM, Sanne I, Scott NA, Shenje J, Sizemore E, Vernon A, Waja Z, Weiner M, Swindells S, Chaisson RE; AIDS Clinical Trials Group; Tuberculosis Trials Consortium. Four-Month Rifapentine Regimens with or without Moxifloxacin for Tuberculosis. N Engl J Med. 2021 May 6;384(18):1705-1718. doi: 10.1056/NEJMoa2033400. PMID 33951360
- [Derived] Scott NA, Lee KK, Sadowski C, Kurbatova EV, Goldberg SV, Nsubuga P, Kitshoff R, Whitelaw C, Thuy HN, Batra K, Allen-Blige C, Davis H, Kim J, Phan M, Fedrick P, Chiu KW, Heilig CM, Sizemore E; AIDS Clinical Trials Group and The Tuberculosis Trials Consortium. Optimizing drug inventory management with a web-based information system: The TBTC Study 31/ACTG A5349 experience. Contemp Clin Trials. 2021 Jun;105:106377. doi: 10.1016/j.cct.2021.106377. Epub 2021 Mar 29. PMID 33794353
- [Derived] Bryant KE, Yuan Y, Engle M, Kurbatova EV, Allen-Blige C, Batra K, Brown NE, Chiu KW, Davis H, Elskamp M, Fagley M, Fedrick P, Hedges KNC, Narunsky K, Nassali J, Phan M, Phan H, Purfield AE, Ricaldi JN, Robergeau-Hunt K, Whitworth WC, Sizemore EE; AIDS Clinical Trials Group; Tuberculosis Trials Consortium. Central monitoring in a randomized, open-label, controlled phase 3 clinical trial for a treatment-shortening regimen for pulmonary tuberculosis. Contemp Clin Trials. 2021 May;104:106355. doi: 10.1016/j.cct.2021.106355. Epub 2021 Mar 10. PMID 33713841
- [Derived] Dorman SE, Nahid P, Kurbatova EV, Goldberg SV, Bozeman L, Burman WJ, Chang KC, Chen M, Cotton M, Dooley KE, Engle M, Feng PJ, Fletcher CV, Ha P, Heilig CM, Johnson JL, Lessem E, Metchock B, Miro JM, Nhung NV, Pettit AC, Phillips PPJ, Podany AT, Purfield AE, Robergeau K, Samaneka W, Scott NA, Sizemore E, Vernon A, Weiner M, Swindells S, Chaisson RE; AIDS Clinical Trials Group and the Tuberculosis Trials Consortium. High-dose rifapentine with or without moxifloxacin for shortening treatment of pulmonary tuberculosis: Study protocol for TBTC study 31/ACTG A5349 phase 3 clinical trial. Contemp Clin Trials. 2020 Mar;90:105938. doi: 10.1016/j.cct.2020.105938. Epub 2020 Jan 22. PMID 31981713

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 34 clinical research sites in 13 countries between January 2016 and October 2018. First participant was enrolled on 25 January 2016. Last participant was enrolled on 30 October 2018.
Pre-assignment Details: Of 5214 participants screened, 2049 did not meet the eligible criteria, 405 declined to participate and site decided not to enroll 145 participants. 2516 participants were randomized Participants were required to have at least one sputum specimen positive for acid-fast bacilli by smear microscopy or positive for M. tuberculosis by Xpert MTB/RIF testing with semiquantitative result of medium or highand susceptible to isoniazid, rifampin, and fluoroquinolones
Groups:
- Regimen 1 (2HRZE/4HR): Eight weeks of daily treatment with rifampin, isoniazid, pyrazinamide, and ethambutol, followed by Eighteen weeks of daily treatment with rifampin and isoniazid
  All drugs are administered orally, seven days/week, directly observed by a health care worker at least five of the seven days each week. Pyridoxine (vitamin B6), 25 or 50 mg, is administered with each study dose. Study drug doses: rifampin, 600 mg; isoniazid, 300 mg; pyrazinamide, < 55kg 1000 mg, >= 55-75 kg 1500 mg, >75 kg 2000 mg; ethambutol, < 55kg 800 mg, >= 55-75 kg 1200 mg, >75 kg 1600 mg
  study drug doses: rifampin, 600 mg; isoniazid, 300 mg; pyrazinamide, < 55kg 1000 mg, >= 55-75 kg 1500 mg, >75 kg 2000 mg; ethambutol, < 55kg 800 mg, >= 55-75 kg 1200 mg, >75 kg 1600 mg
  control: standard six-month treatment
- Regimen 2 (2HPZ/2HP): Eight weeks of daily treatment with rifapentine, isoniazid, pyrazinamide, and ethambutol, followed by Nine weeks of daily treatment with rifapentine and isoniazid
  All drugs are administered orally, seven days/week, directly observed by a health care worker at least five of the seven days each week. Pyridoxine (vitamin B6), 25 or 50 mg, is administered with each study dose. Study drug doses: rifapentine 1200 mg; isoniazid, 300 mg; pyrazinamide, < 55kg 1000 mg, >= 55-75 kg 1500 mg, >75 kg 2000 mg; ethambutol, < 55kg 800 mg, >= 55-75 kg 1200 mg, >75 kg 1600 mg
  study drug doses: rifapentine 1200 mg; isoniazid, 300 mg; pyrazinamide, < 55kg 1000 mg, >= 55-75 kg 1500 mg, >75 kg 2000 mg; ethambutol, < 55kg 800 mg, >= 55-75 kg 1200 mg, >75 kg 1600 mg
  rifapentine: Regimen 2: Rifapentine is substituted for rifampin as the basis of 4-month treatment
- Regimen 3 (2HPMZ/2HPM): Eight weeks of daily treatment with rifapentine, isoniazid, pyrazinamide, and moxifloxacin, followed by Nine weeks of daily treatment with rifapentine, isoniazid, and moxifloxacin
  All drugs are administered orally, seven days/week, directly observed by a health care worker at least five of the seven days each week. Pyridoxine (vitamin B6), 25 or 50 mg, is administered with each study dose. Study drug doses: rifapentine 1200 mg; isoniazid, 300 mg; pyrazinamide, < 55kg 1000 mg, >= 55-75 kg 1500 mg, >75 kg 2000 mg; ethambutol, < 55kg 800 mg, >= 55-75 kg 1200 mg, >75 kg 1600 mg
  study drug doses: rifapentine 1200 mg; isoniazid, 300 mg; pyrazinamide, < 55kg 1000 mg, >= 55-75 kg 1500 mg, >75 kg 2000 mg; moxifloxacin, 400 mg
  rifapentine and moxifloxacin: Regimen 3: In addition to the single substitution described for regimen 2, a second substitution is added, of moxifloxacin for ethambutol.
Period: Overall Study
Arm/Group | Regimen 1 (2HRZE/4HR) | Regimen 2 (2HPZ/2HP) | Regimen 3 (2HPMZ/2HPM)
Started | 829 | 838 | 849
Microbiologically Eligible Analysis Population (Microbiologically Eligible Population included all enrolled participants that received a treatment assignment but excluded the participants with no evidence of cultures positive for M. tuberculosis, or with resistance to one or more of isoniazid, rifampin or fluoroquinolones, or are enrolled in violation of eligibility criteria) | 768 | 784 | 791
Assessable Population (Excluded the Microbiologically eligible participants without an assessable outcome (if they were not already classified as unfavorable and additionally did not attend12M visit but were culture negative when last seen, or had treatment changed due to pregnancy, or died during follow-up with cause unrelated to tuberculosis, or received additional treatment for tuberculosis following exogenous reinfection shown by whole genome sequencing, or died from a violent or accidental death during treatment) | 726 | 752 | 756
Completed (Completed Population included all participants that are randomized and are microbiologically eligible with an Assessable outcome (Assessable Population)) | 726 | 752 | 756
Not Completed | 103 | 86 | 93
Not completed — Death | 3 | 4 | 8
Not completed — Lost to Follow-up | 31 | 23 | 22
Not completed — Pregnancy | 8 | 4 | 5
Not completed — Protocol Violation | 8 | 8 | 4
Not completed — Baseline Drug Resistance | 49 | 40 | 51
Not completed — No positive Mycobacterium tuberculosis culture | 4 | 6 | 3
Not completed — Reinfection with a new strain of MTB | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Population Description: The population is the Microbiologically eligible population that included the randomized participants excluding the ones with no evidence of cultures positive for M. tuberculosis, or with resistance to one or more of isoniazid, rifampin or fluoroquinolones, or are enrolled in violation of eligibility criteria
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen 1 (2HRZE/4HR) | Regimen 2 (2HPZ/2HP) | Regimen 3 (2HPMZ/2HPM) | Total
Number analyzed (Participants) | 768 | 784 | 791 | 2343
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19 | 19 | 25 | 63
  Between 18 and 65 years | 743 | 755 | 755 | 2253
  >=65 years | 6 | 10 | 11 | 27
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30.9 [24.9 to 41.0] | 31.0 [24.6 to 41.1] | 31.0 [24.6 to 41.5] | 31.0 [24.6 to 41.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 224 | 221 | 228 | 673
  Male | 544 | 563 | 563 | 1670
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 20 | 27 | 74
  Not Hispanic or Latino | 287 | 283 | 297 | 867
  Unknown or Not Reported | 454 | 481 | 467 | 1402
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 86 | 93 | 89 | 268
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 553 | 571 | 552 | 1676
  White | 15 | 8 | 13 | 36
  More than one race | 111 | 111 | 135 | 357
  Unknown or Not Reported | 3 | 1 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 7 | 10 | 25
  Africa | 565 | 573 | 578 | 1716
  South Asia | 86 | 89 | 88 | 263
  South America | 109 | 115 | 115 | 339
HIV Status [Count of Participants; unit: Participants] — Randomization was stratified by the presence of cavitation on chest radiograph at baseline (since cavitation is associated with a decreased rate of microbiological response to TB treatment) and by HIV status (HIV-uninfected vs. HIV-infected).
  Participants
    HIV Negative | 704 | 716 | 729 | 2149
    HIV Positive | 64 | 68 | 62 | 194
Cavitation status at Baseline [Count of Participants; unit: Participants]
  Cavitation on chest radiograph | 558 | 573 | 572 | 1703
  No cavitation on chest radiograph | 204 | 205 | 210 | 619
  Unknown | 6 | 6 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: TB Disease-free Survival at 12M After Study Treatment Assignment Among Participants in Control Regimen, Regimen1 (2HRZE/4HR) to Experimental Regimens, Regimen3 (2HPZM/2HPM) and Regimen2 (2HPZ/2HP) (Modified Intent to Treat [MITT] Population)
Description: To evaluate the efficacy of a rifapentine-containing regimen to determine whether the single substitution of rifapentine for rifampin makes it possible to reduce to seventeen weeks the duration of treatment for drug-susceptible pulmonary tuberculosis To evaluate the efficacy of a rifapentine-containing regimen that in addition substitutes moxifloxacin for ethambutol and continues moxifloxacin during the continuation phase, to determine whether it is possible to reduce to seventeen weeks the duration of treatment for drug-susceptible pulmonary tuberculosis A primary outcome status of "favorable", "unfavorable", or "not assessable" was assigned. For detailed definitions of outcomes please refer to: Dorman SE, at al. N Engl J Med. 2021 May 6;384(18):1705-1718.
Time Frame: Twelve months after treatment assignment
Population: The population is the Microbiologically eligible population that included the randomized participants excluding the ones with no evidence of cultures positive for M. tuberculosis, or with resistance to one or more of isoniazid, rifampin or fluoroquinolones, or are enrolled in violation of eligibility criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen 1 (2HRZE/4HR) | Regimen 2 (2HPZ/2HP) | Regimen 3 (2HPMZ/2HPM)
Number analyzed (Participants) | 768 | 784 | 791
Participants
  Favorable Outcome | 656 | 645 | 668
  Unfavorable Outcome | 112 | 139 | 123
Statistical Analysis 1: Comparison: Regimen 1 (2HRZE/4HR) vs Regimen 3 (2HPMZ/2HPM); For primary efficacy endpoint, unfavorable outcomes for Arm1(control) vs Arm3(2PHZM/2PHM) will be considered first, if non-inferiority criteria are met, then Arm 1 vs Arm 2(2PHZE/2PH) will be compared. The proportion of participants with unfavorable outcome can be estimated as: if r_a and r_b are the proportions of unfavorable outcome for the two study arms (a=Arm1 and b = Arm2 or Arm3) and if δ is the non-inferiority margin (=6.6%), statistical hypothesis is H_0:r_b-r_a≥δ vs.H_1:r_b-r_a<δ; Test type: Non-Inferiority — Non-inferiority was assessed using the upper bound of the two-sided 95% CI for the difference between the percentage of patients who are classified as having an unfavorable status on the control regimen (2HRZE/ 4 HR) and the investigational regimens, Regimen 2 (2HPZ/2HP) and Regimen 3 (2HPZM/2HPM). If the upper bound of the confidence interval is less than , then the non-inferiority of Arm 2 or Arm 3 to Arm 1 with a significance level of 0.05 is established (equivalent to one-sided α=0.025); p = 0.05, Cochran-Mantel-Haenszel — For a significance level of 0.05, the statistical test is equivalent to obtaining the two-sided 95% confidence interval for the difference of r_b-r_a; Risk Difference (RD) = 1, 95% CI 2-sided [-2.6 to 4.5]
Statistical Analysis 2: Comparison: Regimen 1 (2HRZE/4HR) vs Regimen 3 (2HPMZ/2HPM); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.05, Cochran-Mantel-Haenszel; For a significance level of 0.05, the statistical test is equivalent to obtaining the two-sided 95% confidence interval for the difference of r_b-r_a; Risk Difference (RD) = 3, 95% CI 2-sided [-0.6 to 6.6]

2. Primary Outcome: TB Disease-free Survival at 12M After Study Treatment Assignment Among Participants in Control Regimen, Regimen1 (2HRZE/4HR) to Experimental Regimens, Regimen3 (2HPZM/2HPM) and Regimen2 (2HPZ/2HP) (Assessable Population)
Description: * To evaluate the efficacy of a rifapentine-containing regimen to determine whether the single substitution of rifapentine for rifampin makes it possible to reduce to seventeen weeks the duration of treatment for drug-susceptible pulmonary tuberculosis
  * To evaluate the efficacy of a rifapentine-containing regimen that in addition substitutes moxifloxacin for ethambutol and continues moxifloxacin during the continuation phase, to determine whether it is possible to reduce to seventeen weeks the duration of treatment for drug-susceptible pulmonary tuberculosis A primary outcome status of "favorable", "unfavorable", or "not assessable" was assigned. For detailed definitions of outcomes please refer to: Dorman SE, at al. N Engl J Med. 2021 May 6;384(18):1705-1718.
Time Frame: Twelve months after treatment assignment
Population: Excluded Microbiologically eligible participants without an assessable outcomes, if they were not already classified as unfavorable and also did not attend 12M visit but were culture negative when last seen, or had treatment changed due to pregnancy, or died during follow-up with cause unrelated to tuberculosis, or received additional treatment for tuberculosis following exogenous reinfection demonstrated by whole genome sequencing, or died from a violent or accidental death during treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen 1 (2HRZE/4HR) | Regimen 2 (2HPZ/2HP) | Regimen 3 (2HPMZ/2HPM)
Number analyzed (Participants) | 726 | 752 | 756
Participants
  Favorable | 656 | 645 | 668
  Unfavorable | 70 | 107 | 88
Statistical Analysis 1: Comparison: Regimen 1 (2HRZE/4HR) vs Regimen 3 (2HPMZ/2HPM); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.05, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 2, 95% CI 2-sided [-1.1 to 5.1]
Statistical Analysis 2: Comparison: Regimen 1 (2HRZE/4HR) vs Regimen 2 (2HPZ/2HP); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.05, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 4.4, 95% CI 2-sided [1.2 to 7.7]

3. Primary Outcome: Percentage Participants With Grade 3 or Higher Adverse Events During Study Drug Treatment in Control Regimen (Regimen 1 2HRZE/4HR) Compared to Experimental Regimens, Regimen 3 (2HPZM/2HPM) and Regimen 2 (2HPZ/2HP) (Safety Analysis Population)
Description: * To evaluate the Safety of a rifapentine-containing regimen to determine whether the single substitution of rifapentine for rifampin makes it possible to reduce to seventeen weeks the duration of treatment for drug-susceptible pulmonary tuberculosis
  * To evaluate the Safety of a rifapentine-containing regimen that in addition substitutes moxifloxacin for ethambutol and continues moxifloxacin during the continuation phase, to determine whether it is possible to reduce to seventeen weeks the duration of treatment for drug-susceptible pulmonary tuberculosis Grade 3 or higher Adverse Events are collected by Clinical sites in systematic way through the laboratory tests and physical exam during regular study follow up visits and also in a non-systematic way when it was self-reported by participants during the study visits. The events are graded by site investigators per Common Terminology Criteria for Adverse Events (CTCAE V4.03
Time Frame: Four months and up to 14 days after last does of after study treatment (Regimen 2 and 3) or Six months and up to 14 days after last does of after study treatment (Regimen 1)
Population: Safety analyses included all randomized participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen 1 (2HRZE/4HR) | Regimen 2 (2HPZ/2HP) | Regimen 3 (2HPMZ/2HPM)
Number analyzed (Participants) | 825 | 835 | 846
Participants
  Participants with Grade 3 or higher Adverse events | 159 | 119 | 159
  Participants with less than Grade 3 Adverse Events or no adverse events | 666 | 716 | 687
Statistical Analysis 1: Comparison: Regimen 1 (2HRZE/4HR) vs Regimen 3 (2HPMZ/2HPM); For primary Safety endpoint, unfavorable outcomes for Arm1(control) vs Arm3(2PHZM/2PHM) will be considered first, if non-inferiority criteria are met, then Arm 1 vs Arm 2(2PHZE/2PH) will be compared. The proportion of participants with unfavorable outcome can be estimated as: if r_a and r_b are the proportions of unfavorable outcome for the two study arms (a=Arm1 and b = Arm2 or Arm3) and if δ is the non-inferiority margin (=6.6%), statistical hypothesis is H_0:r_b-r_a≥δ vs.H_1:r_b-r_a<δ; Test type: Non-Inferiority — Non-inferiority was assessed using the upper bound of the two-sided 95% CI for the difference between the percentage of patients who are classified as having an unfavorable status on the control regimen (2HRZE/ 4 HR) and the investigational regimens, Regimen 2 (2HPZ/2HP) and Regimen 3 (2HPZM/2HPM). If the upper bound of the confidence interval is less than, then the non-inferiority of Arm 2 or Arm 3 to Arm 1 with a significance level of 0.05 is established (equivalent to one-sided α=0.025); p = 0.05, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = -0.6, 95% CI 2-sided [-4.3 to 3.2]
Statistical Analysis 2: Comparison: Regimen 1 (2HRZE/4HR) vs Regimen 2 (2HPZ/2HP); [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.05, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = -5.1, 95% CI 2-sided [-8.7 to -1.5]

4. Secondary Outcome: Proportion of Participants Who Are Culture Negative at Eight Weeks
Description: Proportion of participants who are culture negative at eight weeks, liquid media
Time Frame: eight weeks
Population: Microbiologically eligible analysis population, evaluable patients (positive or negative culture result)
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen 1 (2HRZE/4HR) | Regimen 2 (2HPZ/2HP) | Regimen 3 (2HPMZ/2HPM)
Number analyzed (Participants) | 682 | 704 | 698
Participants | 523 | 616 | 641

5. Secondary Outcome: Time to Stable Sputum Culture Conversion
Description: Time to stable sputum culture conversion, liquid media
Time Frame: four or six months
Population: Microbiologically Eligible Analysis Population
Measure: Median (Inter-Quartile Range); unit: weeks
Groups:
- Regimen 1: Eight weeks of daily treatment with rifampin, isoniazid, pyrazinamide, and ethambutol, followed by Eighteen weeks of daily treatment with rifampin and isoniazid
  All drugs are administered orally, seven days/week, directly observed by a health care worker at least five of the seven days each week. Pyridoxine (vitamin B6), 25 or 50 mg, is administered with each study dose.
  study drug doses: rifampin, 600 mg; isoniazid, 300 mg; pyrazinamide, < 55kg 1000 mg, >= 55-75 kg 1500 mg, >75 kg 2000 mg; ethambutol, < 55kg 800 mg, >= 55-75 kg 1200 mg, >75 kg 1600 mg
  control: standard six-month treatment
- Regimen 2: Eight weeks of daily treatment with rifapentine, isoniazid, pyrazinamide, and ethambutol, followed by Nine weeks of daily treatment with rifapentine and isoniazid
  All drugs are administered orally, seven days/week, directly observed by a health care worker at least five of the seven days each week. Pyridoxine (vitamin B6), 25 or 50 mg, is administered with each study dose.
  study drug doses: rifapentine 1200 mg; isoniazid, 300 mg; pyrazinamide, < 55kg 1000 mg, >= 55-75 kg 1500 mg, >75 kg 2000 mg; ethambutol, < 55kg 800 mg, >= 55-75 kg 1200 mg, >75 kg 1600 mg
  rifapentine: Regimen 2: Rifapentine is substituted for rifampin as the basis of 4-month treatment
- Regimen 3: Eight weeks of daily treatment with rifapentine, isoniazid, pyrazinamide, and moxifloxacin, followed by Nine weeks of daily treatment with rifapentine, isoniazid, and moxifloxacin
  All drugs are administered orally, seven days/week, directly observed by a health care worker at least five of the seven days each week. Pyridoxine (vitamin B6), 25 or 50 mg, is administered with each study dose.
  study drug doses: rifapentine 1200 mg; isoniazid, 300 mg; pyrazinamide, < 55kg 1000 mg, >= 55-75 kg 1500 mg, >75 kg 2000 mg; moxifloxacin, 400 mg
  rifapentine and moxifloxacin: Regimen 3: In addition to the single substitution described for regimen 2, a second substitution is added, of moxifloxacin for ethambutol.
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3
Number analyzed (Participants) | 768 | 784 | 791
weeks | 8.14 [8.00 to 12.14] | 8.14 [4.14 to 12.00] | 8.14 [4.14 to 8.29]

6. Secondary Outcome: Discontinuation of Assigned Treatment for a Reason Other Than Microbiological Ineligibility (Tolerability)
Description: Tolerability of the regimen is evaluated using the outcome of discontinuation of assigned treatment for a reason other than microbiological ineligibility.
Time Frame: four or six months
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen 1 (2HRZE/4HR) | Regimen 2 (2HPZ/2HP) | Regimen 3 (2HPMZ/2HPM)
Number analyzed (Participants) | 825 | 835 | 846
Participants | 61 | 37 | 55

7. Secondary Outcome: Estimated Steady State Efavirenz PK Parameters Including Mid-dosing Interval Concentration
Description: Among participants with HIV infection receiving efavirenz-based antiretroviral therapy, number of participants who maintained plasma efavirenz concentrations ≥1 mg/L during TB treatment.
Time Frame: four months
Population: Analysis Population Description: This analysis population includes participants in EFV group 1 who were already on an EFV-containing ART regimen when initiating RPT-based TB treatment (experimental arms only). That is, this analysis was pre-specified to report data by pooling participants from Regimen 2 (2HPZE/2HP) and Regimen 3 (2HPMZ/2HPM) who were on an EFV-containing ART regimen.
Measure: Count of Participants; unit: Participants
Groups:
- EFV1: Individuals with HIV already receiving an efavirenz based ART regimen and randomized to one of the rifapentine based treatment arms of the study (efavirenz group 1, EFV1).
Arm/Group | EFV1
Number analyzed (Participants) | 67
Participants | 62

8. Secondary Outcome: TB Disease-free Survival at Eighteen Months After Study Treatment Assignment
Description: * To evaluate the efficacy of a rifapentine-containing regimen to determine whether the single substitution of rifapentine for rifampin makes it possible to reduce to seventeen weeks the duration of treatment for drug-susceptible pulmonary tuberculosis
  * To evaluate the efficacy of a rifapentine-containing regimen that in addition substitutes moxifloxacin for ethambutol and continues moxifloxacin during the continuation phase, to determine whether it is possible to reduce to seventeen weeks the duration of treatment for drug-susceptible pulmonary tuberculosis
Time Frame: Eighteen months after study treatment assignment.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen 1 (2HRZE/4HR) | Regimen 2 (2HPZ/2HP) | Regimen 3 (2HPMZ/2HPM)
Number analyzed (Participants) | 768 | 784 | 791
Participants
  Favorable | 656 | 636 | 667
  Unfavorable | 112 | 148 | 124
Statistical Analysis 1: Comparison: Regimen 1 (2HRZE/4HR) vs Regimen 3 (2HPMZ/2HPM); Test type: Non-Inferiority — Margin to define inferiority: 6.6% (δ = 0.066); Risk Difference (RD) = 1.09, 95% CI 2-sided [-2.45 to 4.63]
Statistical Analysis 2: Comparison: Regimen 1 (2HRZE/4HR) vs Regimen 2 (2HPZ/2HP); Test type: Non-Inferiority — Margin to define inferiority: 6.6% (δ = 0.066); Risk Difference (RD) = 4.12, 95% CI 2-sided [0.45 to 7.79]

9. Secondary Outcome: TB Disease-free Survival at Eighteen Months After Study Treatment Assignment
Description: as for outcome 8
Time Frame: Eighteen months after treatment assignment
Population: Assessable Population: Excluded the Microbiologically eligible pts without an assessable outcomes as if they were not already classified as unfavorable and add did not attend mo12 visit but were culture negative when last seen, or had treatment changed due to pregnancy, or died during follow-up with cause unrelated to tuberculosis, or received additional treatment for tuberculosis following exogenous reinfection demonstrated by WGS, or died from a violent or accidental death during treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen 1 (2HRZE/4HR) | Regimen 2 (2HPZ/2HP) | Regimen 3 (2HPMZ/2HPM)
Number analyzed (Participants) | 725 | 733 | 746
Participants
  Favorable | 656 | 636 | 667
  Unfavorable | 69 | 97 | 79
Statistical Analysis 1: Comparison: Regimen 1 (2HRZE/4HR) vs Regimen 3 (2HPMZ/2HPM); Test type: Non-Inferiority — Margin to define inferiority: 6.6% (δ = 0.066); Risk Difference (RD) = 1.05, 95% CI 2-sided [-2.01 to 4.11]
Statistical Analysis 2: Comparison: Regimen 1 (2HRZE/4HR) vs Regimen 2 (2HPZ/2HP); Test type: Non-Inferiority — Margin to define inferiority: 6.6% (δ = 0.066); Risk Difference (RD) = 3.66, 95% CI 2-sided [0.42 to 6.90]

10. Secondary Outcome: Speed of Decline of Sputum Viable Bacilli by Automated Liquid MGIT Culture Days to Detection
Description: Parameter estimates of the nonlinear mixed effect models describing longitudinal time to positive (TTP)
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: log10 DTP / day
Arm/Group | Regimen 1 (2HRZE/4HR) | Regimen 2 (2HPZ/2HP) | Regimen 3 (2HPMZ/2HPM)
Number analyzed (Participants) | 768 | 784 | 791
log10 DTP / day | 0.14 | 0.20 | 0.24

11. Other Pre Specified Outcome: Sensitivity Analyses Assuming All Losses to Follow-up and Non-tuberculosis Deaths Have an Unfavorable Outcome
Description: A sensitivity analysis used to supplement the primary efficacy results and provide further insight into whether the intervention regimens should be considered to have non-inferior efficacy. This analysis considers the difference in proportion of unfavorable outcomes between the control arm and each of the experimental arms.
  Measurement Description: The difference in proportion unfavorable was calculated using a stratified analysis using Cochran-Mantel-Haenszel weights. The analysis was stratified by HIV status and presence of cavitation only, and the stratified difference was considered primary.
Time Frame: 12 months
Population: Microbiologically eligible analysis population.
Measure: Count of Participants; unit: Participants
Groups:
- Regimen 2 (2HPEZ/2HP): Eight weeks of daily treatment with rifapentine, isoniazid, pyrazinamide, and ethambutol, followed by Nine weeks of daily treatment with rifapentine and isoniazid
  All drugs are administered orally, seven days/week, directly observed by a health care worker at least five of the seven days each week. Pyridoxine (vitamin B6), 25 or 50 mg, is administered with each study dose. Study drug doses: rifapentine 1200 mg; isoniazid, 300 mg; pyrazinamide, < 55kg 1000 mg, >= 55-75 kg 1500 mg, >75 kg 2000 mg; ethambutol, < 55kg 800 mg, >= 55-75 kg 1200 mg, >75 kg 1600 mg
  study drug doses: rifapentine 1200 mg; isoniazid, 300 mg; pyrazinamide, < 55kg 1000 mg, >= 55-75 kg 1500 mg, >75 kg 2000 mg; ethambutol, < 55kg 800 mg, >= 55-75 kg 1200 mg, >75 kg 1600 mg
  rifapentine: Regimen 2: Rifapentine is substituted for rifampin as the basis of 4-month treatment
Arm/Group | Regimen 1 (2HRZE/4HR) | Regimen 2 (2HPEZ/2HP) | Regimen 3 (2HPMZ/2HPM)
Number analyzed (Participants) | 768 | 784 | 791
Participants | 656 | 645 | 668
Statistical Analysis 1: Comparison: Regimen 1 (2HRZE/4HR) vs Regimen 2 (2HPEZ/2HP); Test type: Non-Inferiority — Margin to define inferiority: 6.6% (δ = 0.066); Risk Difference (RD) = 3.0, 95% CI 2-sided [-0.6 to 6.6]
Statistical Analysis 2: Comparison: Regimen 1 (2HRZE/4HR) vs Regimen 3 (2HPMZ/2HPM); Test type: Non-Inferiority — Margin to define inferiority: 6.6% (δ = 0.066); Risk Difference (RD) = 2.29, 95% CI 2-sided [-1.12 to 5.70]

12. Other Pre Specified Outcome: Sensitivity Analyses Assuming All Losses to Follow-up and Non-tuberculosis Deaths Have a Favorable Outcome
Description: as for outcome 11
Time Frame: 12 months
Population: Assessable analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen 1 (2HRZE/4HR) | Regimen 2 (2HPEZ/2HP) | Regimen 3 (2HPMZ/2HPM)
Number analyzed (Participants) | 726 | 752 | 756
Participants | 671 | 650 | 673
Statistical Analysis 1: Comparison: Regimen 1 (2HRZE/4HR) vs Regimen 2 (2HPEZ/2HP); Test type: Non-Inferiority — Margin to define inferiority: 6.6% (δ = 0.066); Risk Difference (RD) = 5.9, 95% CI 2-sided [2.8 to 8.9]
Statistical Analysis 2: Comparison: Regimen 1 (2HRZE/4HR) vs Regimen 3 (2HPMZ/2HPM); Test type: Non-Inferiority — Margin to define inferiority: 6.6% (δ = 0.066); Risk Difference (RD) = 3.4, 95% CI 2-sided [0.5 to 6.3]

ADVERSE EVENTS:
Time Frame: Adverse Events were reported from randomization to up to 14 days after last dose of study treatment Regimen (4 months and up to 14 days or 6 months and up to 14 days); All cause Mortality is reported during study treatment and up to M18 study follow up visit (18 months)
Description: The Safety analysis population included all the randomized patients and received at least 1 dose of trial medication. Grade 3 or higher Adverse Events per CTCAE V4.03 are collected in systematic way through the laboratory tests and physical exam at regular study visits and also non-systematic way when self-reported by participants. All Cause Mortality is adjusted to reflect the deaths occurred up to M18 study visit.
Arm/Group | Regimen 1 (2HRZE/4HR) | Regimen 2 (2HPZ/2HP) | Regimen 3 (2HPMZ/2HPM)
All-Cause Mortality (participants affected / at risk) | 12/825 | 11/835 | 13/846
Serious Adverse Events (participants affected / at risk) | 56/825 | 39/835 | 37/846
Other Adverse Events (participants affected / at risk) | 74/825 | 61/835 | 94/846
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen 1 (2HRZE/4HR) (N=825) | Regimen 2 (2HPZ/2HP) (N=835) | Regimen 3 (2HPMZ/2HPM) (N=846)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 2 (2)
Thrombotic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Myocardial Ischemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Right Ventricular Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic Retinopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumatosis Intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1) | 0 (0)
Drug Intolerance (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 10 (10) | 5 (5) | 7 (7)
Bone Tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dengue Fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Extrapulmonary Tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hepatitis C (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Paracoccidioidal Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
Pneumonia Bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Alcohol Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Chest Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Documented Hypersensitivity To Administered Product (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hand Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Stab Wound (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Traumatic Hemothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT Prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1)
Diabetes Mellitus, Inadequate Control (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sacroilitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Anogenital Warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Neoplasm, Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Esophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous Cell Carcinoma of Tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Central Nervous System Lesion (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Cerebral Infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Guillian-Barre Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Temporal Lobe Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Complication of Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Pre-Eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 3 (3) | 2 (2)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Renal Impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal Tubular Necrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 4 (5) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Drug Reaction with Eosinophilia and Systemic Symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash Generalized (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rash, Maculopapular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3)
Aortic Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 3 (3) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen 1 (2HRZE/4HR) (N=825) | Regimen 2 (2HPZ/2HP) (N=835) | Regimen 3 (2HPMZ/2HPM) (N=846)
Neutropenia (Blood and lymphatic system disorders) | 48 (51) | 34 (39) | 56 (57)
Hepatitis (Hepatobiliary disorders) | 26 (31) | 27 (31) | 38 (40)

LIMITATIONS AND CAVEATS:
A study limitation is that placebos were not used, and therefore neither participants nor site staff were blinded to treatment assignment. Another limitation is that only 8% of participants were HIV-coinfected, limiting the power to compare regimens in this important population

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/72/NCT02410772/Prot_SAP_000.pdf